CLINICAL TRIAL: NCT05626998
Title: The Effect of Intramuscular Dexmedetomidine Versus Oral Gabapentin Premedication on the Emergence Agitation After Rhinoplasty. A Prospective, Randomized, Double-blind Controlled Trial.
Brief Title: Dexmedetomidine Versus Gabapentin Premedication on the Emergence Agitation After Rhinoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tamer Samir Abdelsalam, lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R 164/ 2022
Record Dates: First submitted 2022-11-08; First posted 2022-11-25 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The participants will not receive premedication
- Dexmedetomidine (Active Comparator): The participants will receive intramuscular dexmedetomidine injection (1 µg/kg) diluted in 2ml normal saline thirty minutes before surgery in the ward
  Interventions: Drug: Dexmedetomidine
- Gabapentin (Active Comparator): The participants will receive 600 mg gabapentin (two capsules each containing 300 mg) thirty minutes before surgery in the ward
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Dexmedetomidine — The participants will receive intramuscular dexmedetomidine injection (1 µg/kg) diluted in 2ml normal saline thirty minutes before surgery in the ward.
  Arms: Dexmedetomidine
Drug: Gabapentin — The participants will receive 600 mg gabapentin (two capsules each containing 300 mg) thirty minutes before surgery in the ward
  Arms: Gabapentin

SUMMARY:
To compare the effect of intramuscular dexmedetomidine versus oral gabapentin premedication on the emergence agitation after rhinoplasty.

DETAILED DESCRIPTION:
Emergence agitation (EA) is a clinical condition characterized by agitation, confusion, disorientation, and aggressive behavior in the early phase of recovery from general anesthesia (incidence about 21.3%). This may lead to various injuries, self-extubation, bleeding, increased pain, removal of catheters, increased blood pressure, heart rate, and myocardial oxygen consumption. Premedication with dexmedetomidine and gabapentin are promising options for EA.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade I or II.
* Sex: Both sexes.
* Age between 18 and 40 years.
* Patients scheduled for rhinoplasty under general anesthesia

Exclusion Criteria:

* Declining to give written informed consent.
* History of allergy to the medications used in the study.
* history of cardiovascular diseases including bradycardia, heart block, and hypertension.
* History of chest problems including bronchial asthma.
* Had a history of drug or alcohol abuse.
* Taking opioids or sedative medications.
* Inability to communicate with patients to evaluate postoperative pain.
* Hepatic or renal failure.
* Psychiatric disorders with antipsychotics or antidepressants.
* Bleeding disorders, antiplatelets (aspirin, clopidogrel), or anticoagulant (warfarin).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
emergence agitation (EA) | During first hour of recovery.
  in the form of Riker Sedation-Agitation Scale (where 1 = "unarousable" and 7 = "dangerous agitation" with score ≥5 considered EA).

SECONDARY OUTCOMES:
Postoperative pain in the form of visual analog scale | every 4 hours for 12 hours
  (VAS, 0=no pain; 10=worst possible pain)
Incidence of the common adverse effects | at 12 hours
  nausea and vomiting, dizziness, and headache

CONTACTS AND LOCATIONS:
Overall Officials: tamer S abdelaziz, MD, Principal Investigator — Faculty of medicine, Ain Shams University, Cairo, Egypt
Locations (1):
- faculty of medicine, Ain Shams University, Cairo, Egypt

REFERENCES:
- [Derived] Abdelaziz TSA, Mohammed Elsayed HE, Kamal Eldin DM, Ibrahim IM. "The effect of intramuscular dexmedetomidine versus oral gabapentin premedication on the emergence agitation after rhinoplasty". A prospective, randomized, double-blind controlled trial. BMC Anesthesiol. 2025 Jan 31;25(1):50. doi: 10.1186/s12871-025-02914-5. PMID 39891093